CLINICAL TRIAL: NCT02157701
Title: Polyherbal Capsule Formulation for Joint Health: a Multicenter, 2-arm, Randomized, Double-blind, Placebo-controlled Study
Brief Title: Polyherbal Capsule Formulation for Joint Health
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NewChapter, Inc. (Industry)
Collaborators: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: NEWC2600; 2014020 (Other: Sponsor)
Record Dates: First submitted 2014-06-04; First posted 2014-06-06 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Knee Discomfort; Pain Physical Activity
Keywords: Dietary herbs; Polyherbal capsule; Functional exercise capacity; Joint health

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Polyherbal capsule (Experimental): 1 capsule taken with breakfast and 1 capsule with lunch. Capsules should be taken immediately prior to meals and not with carbonated beverages.
  Interventions: Dietary Supplement: Polyherbal capsule
- Placebo capsule (Placebo Comparator): 1 capsule taken with breakfast and 1 capsule with lunch. Capsules should be taken immediately prior to meals and not with carbonated beverages.
  Interventions: Dietary Supplement: Placebo capsule

INTERVENTIONS:
Dietary Supplement: Polyherbal capsule
  Arms: Polyherbal capsule
Dietary Supplement: Placebo capsule
  Arms: Placebo capsule

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, study in subjects with exercise-related knee pain/discomfort to determine the efficacy of a polyherbal capsule compared to placebo capsule in improving exercise capacity and overall parameters of joint health.

DETAILED DESCRIPTION:
Subjects will come to the study site at Visit 1 for screening assessments (which will occur within 14 days before the start of the run-in period) and to answer questions associated with habitual diet, exercise capacity, and level of activity. Those subjects who meet initial inclusion/exclusion criteria will undergo a run-in period of at least 7 days at home to discontinue use of all concurrent dietary supplements. Subjects will then return to the study site at Visit 2 (Baseline; Day 0) for further assessments and those meeting all inclusion/exclusion criteria will be enrolled into the study and randomly assigned to study product.

Approximately 108 subjects (54 per treatment group) will be enrolled in the study. Subjects will be evaluated at Visit 3 (Day 14), Visit 4 (Day 45), Visit 5 (Day 60, phone call), and Visit 6 (Day 90). Exercise capacity (ie, 6-minute timed walk distance test) will be assessed, along with overall knee wellness and joint-related symptoms using WOMAC, PGA, Knee Pain Rating Scale, and rescue medication usage. Safety will be assessed by collecting adverse events (AEs) and clinical laboratory data.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 25 and ≤ 75 years of age with history of joint discomfort in at least 1 knee following daily activities but otherwise healthy
* body mass index (BMI) ≥ 25 and ≤ 40 kg/m2
* sum of ≥ 60 mm (based on 100-mm visual analog scale [VAS]) on the first 2 questions (ie, "How much pain have you had when walking on a flat surface?" "How much pain have you had when going up or down stairs?") of the WOMAC (Section A; Appendix 2)
* females of child bearing potential must agree to use appropriate birth control methods during the entire study period
* agree not to initiate any new exercise or diet programs during the entire study period
* agree not to change their current diet or exercise program, or to use other dietary supplements other than the test product, during the entire study period
* understand the study procedures and sign the forms providing informed consent to participate in the study, and authorize the release of relevant protected health information of the study investigator.

Exclusion Criteria:

* use of NSAIDS during the study (however 81 mg of aspirin daily for cardioprotection is allowed)
* daily use of dietary supplements and herbal supplements beginning at the screening visit and during the study
* subjects with any history of chronic inflammatory disease, immune system disorder or auto-immune disorder including but not limited to the following: AIDS/HIV, ankylosing spondylitis, dermatomyositis, fibromyalgia, Grave's disease, Hashimoto's thyroiditis, lupus, multiple sclerosis, myasthenia gravis, pernicious anemia, systemic vasculitis conditions such as temporal arteritis, primary biliary cirrhosis, psoriasis, Raynaud's syndrome, rheumatoid arthritis, sarcoidosis, scleroderma including the CREST syndrome subset, Sjogren's syndrome, temporal arteritis, inflammatory bowel disease, vitiligo, or chronic infections such as Lyme disease, tuberculosis, endocarditis, and osteomyelitis;
* history of or current diagnosis of gout or pseudogout
* use of any immunosuppressive drugs or biologic products in the last 12 months (including steroids [except for inhaled and topical dose forms])
* antibiotic use, anticoagulants, intra-articular steroids in past 3 months
* intra-articular hyaluronic acid in past 6 months
* subjects with chronic pain syndrome and who are in the judgment of the Investigator unlikely to respond to any therapy (Note that chronic depression and chronic anxiety are known magnifiers of chronic pain syndrome and are also exclusionary. Chronic fatigue syndrome overlaps with the chronic pain domain and is also exclusionary. In addition, fibromyalgia is a central nervous system (CNS) disorder and overlaps with the chronic pain and chronic fatigue domains and is exclusionary as well.)
* any significant GI condition that would potentially interfere with the evaluation of the study product including but not limited to inflammatory bowel disease (ulcerative colitis or Crohn's), history of lap band surgery, history of perforation of the stomach or intestines, or gastroparesis
* clinically significant renal, hepatic, GI, endocrine (including diabetes mellitus), neurologic (particularly balance or neuropathy problems), or hematologic disorders; or chronic obstructive pulmonary disease (COPD), asthma, lung disease, or heart disease that limits exercise capacity (such as peripheral artery disease, ischemic heart disease, heart failure, stroke in the last year, or uncontrolled hypertension [systolic blood pressure over 140 mmHg and/or diastolic above 90 mmHg]) or causes abnormal respiratory or cardiovascular responses during the 6-minute timed walk distance test (such as angina or arrhythmias)
* known allergy or sensitivity to herbal ingredients in the test products, acetaminophen, olive oil, or soy
* history or presence of cancer in the last 5 years (except basal cell carcinoma of skin or in-situ cervical cancer)
* recent history of (within 2 years) alcohol or substance abuse
* participation in a clinical study with exposure to any non-registered drug product within 30 days prior to this study
* individual has a condition the Investigator believes would interfere with his or her ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results or put the person at undue risk, including subjects who are bed or wheelchair-bound or those who have any physical disability which could interfere with their ability to walk or perform the exercise capacity assessments included in this protocol (eg, history of knee or hip joint replacement surgery)
* diabetes not controlled by medication
* untreated or unstable thyroid dysfunction (hyper- or hypo-thyroidism)
* subjects with a significant mental health disorder (bipolar disorder, chronic depression requiring medication, chronic anxiety disorder, obsessive compulsive disorder, or active eating disorders including anorexia nervosa or bulimia)
* subjects with a history of seizures in the last 5 years or dizziness when exercising
* knee arthroscopy in the previous year or surgeries of the lumbar spine, hip, knee, ankle or foot
* surgery scheduled prior to study completion
* pregnant or lactating women
* walk > 575 meters (1886 feet), or have a Knee Pain Rating Scale (Appendix 4) score of < 40 mm on a 100 mm VAS that assesses knee discomfort, after the 6-minute timed walk distance test.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2014-06; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
6-minute Timed Walk Distance Test | Visit 6 (Day 90)
  Subjects will walk up and down a hallway for 6 minutes after being instructed to walk as rapidly as possible within their comfort zone and without causing themselves any pain. Study personnel will time each subject with a stopwatch and measure the total distance travelled in the 6 minutes.

SECONDARY OUTCOMES:
6-minute timed walk distance test | Visits 3 and 4 (Days 14 and 45, respectively)
WOMAC pain questions | Visits 3, 4, and 6 (Days 14, 45, and 90, respectively)
  WOMAC Index is a self-administered questionnaire that assesses 3 dimensions of pain, physical function, and joint stiffness in knee and hip osteoarthritis using a battery of 24 questions. The latest version of the instrument (WOMAC 3.1) in 100-mm VAS format will be used in this clinical study.
Patient Global Assessment (PGA) | Visits 3, 4, and 6 (Days 14, 45, and 90, respectively)
  PGA is a measurement tool to quantify disease activity that asks patients in 100-mm VAS format to rate on a scale how they feel overall.
WOMAC overall score | Visits 3, 4, and 6 (Days 14, 45, and 90, respectively).
WOMAC physical function questions | Visits 3, 4, and 6 (Days 14, 45, and 90, respectively).
WOMAC joint stiffness questions | Visits 3, 4, and 6 (Days 14, 45, and 90, respectively).
Knee Pain Rating Scale | Visits 3, 4, and 6 (Days 14, 45, and 90, respectively).
  A 100-mm VAS Pain Rating Scale will be used to assess knee discomfort after the 6-minute timed walk distance test, where 0 mm = "No Pain" and 100 mm = "Worst Possible Pain".
Rescue medication usage | Visits 3, 4, and 6 (Days 14, 45, and 90, respectively).
  Acetaminophen will be permitted as rescue product during the treatment phase and at the end of the 6 minute timed walk distance test. Subjects will be advised to use rescue product only in case of unbearable pain and to restrict the use to a maximum of 4 tablets (2 g) per day.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Brum, MD, Study Director — Procter and Gamble
Locations (5):
- United States (5):
  - Akta Medika Medical Group Research Division, Homestead, Florida
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Radiant Research, Dallas, Texas
  - Benchmark Research, San Angelo, Texas
  - Radiant Research, San Antonio, Texas